CLINICAL TRIAL: NCT01636908
Title: Pilot Study on the Determination of Intratumoral Concentrations of Kinase Inhibitors in Patients With Advanced Solid Malignancies.
Brief Title: Determination of Intratumoral Concentrations of Kinase Inhibitors in Patients With Advanced Solid Malignancies.
Acronym: ICK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, M. Labots, Medical Oncologist, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011/128
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Cancer; Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — Sunitinib; Sorafenib; Erlotinib Hydrochloride; Everolimus; Lapatinib; Dasatinib; pazopanib; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kinase inhibitor (Experimental): Patients are cohort-wise treated with a registered (tyrosine) kinase inhibitor
  Interventions: Drug: Sunitinib; Drug: Sorafenib; Drug: Erlotinib; Drug: Everolimus; Drug: Lapatinib; Drug: Dasatinib; Drug: Pazopanib; Drug: Vemurafenib; Procedure: tumor biopsy; Procedure: skin biopsy (optional)

INTERVENTIONS:
Drug: Sunitinib — 50 mg once daily, oral use, 14 days
Drug: Sorafenib — 400 mg, twice daily, oral use, 14 days
Drug: Erlotinib — 150 mg once daily, oral use, 14 days
Drug: Everolimus — 10 mg once daily, oral use, 14 days
Drug: Lapatinib — 1250 mg once daily, oral use, 14 days
Drug: Dasatinib — 100 mg once daily, oral use, 14 days
Drug: Pazopanib — 800 mg once daily, oral use, 14 days
Drug: Vemurafenib — 960 mg twice daily, oral use, 15-21 days
Procedure: tumor biopsy
Procedure: skin biopsy (optional)

SUMMARY:
The purpose of this study is to determine intratumoral concentration of kinase inhibitors upon 2 weeks of treatment in tumor tissue of patients.

DETAILED DESCRIPTION:
Patients will be cohort-wise treated with clinically available kinase inhibitors for 2 weeks prior to standard palliative treatment. Five patients will be included in each of eight drug cohorts. Biopsies will be performed to determine intratumoral drug concentrations and to compare tissue (phospho)proteomic and kinase activity profiles before and during therapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid malignancy
* minimum age 18 years
* indication for palliative treatment
* measurable disease with at least one lesion accessable for biopsy

Exclusion Criteria:

* Cardiovascular conditions including congestive heartfailure NYHA class >2
* recent myocardial infarction or uncontrolled coronary artery disease
* cardiac arrhythmias requiring anti-arrhythmic therapy
* uncontrolled hypertension
* uncontrolled infections
* serious non-healing wound, ulcer or bone fracture
* pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
concentrations of intratumoral kinase inhibitors upon 2 weeks of treatment | 2 weeks

SECONDARY OUTCOMES:
kinase inhibitor concentrations in plasma, serum and PBMC's upon 2 weeks of treatment | 2 weeks
intra-dermal kinase inhibitor concentrations upon 2 weeks of treatment | 2 weeks
To determine per patient whether 2 weeks of treatment with kinase inhibitors induces significant change of phosphoproteomic profiles in tumor tissue | 2 weeks
To determine per patient whether 2 weeks of treatment with kinase inhibitors induces significant change of kinase activity in tumor tissue | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: H.M.W. Verheul, MD, PhD, Principal Investigator — VU Medical Center Amsterdam
Locations (1):
- VUMedical Center, Amsterdam, Netherlands